CLINICAL TRIAL: NCT04875832
Title: Eye Movement Desensitization and Reprocessing for Depressed People With Multiple Sclerosis: A Pilot Study
Brief Title: EMDR for Depressed People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: EMDR Europe (Industry); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5_16/10/2019
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis; Depression
Keywords: Multiple Sclerosis; Depression; EMDR; Qualiti of life; MRI
MeSH Terms: conditions — Multiple Sclerosis; Depression | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Pre versus post EMDR treatment feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervetion Group (Experimental): EMDR intervention group
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing - EMDR

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing - EMDR — EMDR is a comprehensive psychotherapy approach, originally developed to treat the victims of trauma. EMDR is guided by an information processing model known as the Adaptive Information Processing (AIP) model. One of the key assumptions of the AIP model is that dysfunctionally stored (disturbing) memories are the cause of several mental pathologies. EMDR is therefore used to address a range of complaints that follow distressing life experiences and it
  is characterized by an eight-phase psychotherapy approach. The intervention is based on the use of bilateral stimulation (e.g., taps, tones, or eye movements), which aims to stimulate the information processing system of the brain in combination with other methods of established psychotherapies. EMDR is widely recognized as an empirically supported treatment for post-traumatic stress disorder (PTSD) and it is one of the best psychological treatment focused on the ri-processing of recent traumatic experiences

SUMMARY:
Several studies have reported high rates of depression in people with MS. Depressive symptoms represent a serious threat to quality of life and well-being. Furthermore, findings from the literature suggest that mechanisms underneath depressive features and loss of physical functions in MS could be related. The current study aims at investigating the feasibility of a fairly new type of psychotherapy known as "eye movement desensitization and reprocessing" (EMDR) on depression in people with MS. The goal of this intervention is to reduce the long-lasting effects of distressing memories by developing more adaptive coping mechanisms, through bilateral sensory stimulation. Together with the study on clinical measures, brain mechanisms of change will be assessed with MRI. Fifteen depressed or mildly depressed people with MS will be recruited. Participants will be assessed for depression, and quality of life, before and after the intervention. Participants will also undergo an MRI for brain structural and functional assessments before and after the EMDR intervention. The main aim of the study is to verify that EMDR is a feasible psychotherapeutic approach for people with depression and MS and to collect preliminary data on the efficacy of this type of intervention in reducing the depressive symptoms and improving the quality of life. The study, however, will not be limited to the analysis of outcome differences. The use of MRI assessments, in fact, will allow to explore possible brain change modifications related to depression reduction and/or symptoms modifications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting or progressive MS.
* Presence of depressive symptomatology, with HADS scores > 8, confirmed by HDRS scores (clinical interview) > 14.
* No change of pharmacological treatment in the 3 months before the enrolment.
* Ability to communicate and to understand tasks.
* No clinical relapses or use of steroid treatment during the 4 weeks before the enrolment.
* Provided informed consent for study participation.

Exclusion Criteria:

* Severe co-morbidity that would reduce life expectancy to less than one year (i.e. end-stage oncological diseases or severe cardiac dysfunction).
* Severe neuropsychological impairment evaluated with the MMSE.
* Psychosis or dissociative disorders.
* No current psychotherapy treatment
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | Change between the baseline (before EMDR treatment-T0), the end of the EMDR intervention lasting three months (T1) and the follow up at three months after the end of the intervention (T2)
  clinical structured interview aimed to evaluate the presence of depressive symptoms
Hospital Anxiety and Depression Scale (HADS) | Change between the baseline (before EMDR treatment-T0), the end of the EMDR intervention lasting three months (T1) and the follow up at three months after the end of the intervention (T2)
  A self-report assessment for anxious and depressive symptoms

SECONDARY OUTCOMES:
Multiple Scleroris Quality of Life - 54, MSQoL-54 | Change between the baseline (before EMDR treatment-T0), the end of the EMDR intervention lasting three months (T1) and the follow up at three months after the end of the intervention (T2)
  A multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. It is composed by 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function.
Brain MRI | Change between the baseline (before EMDR treatment-T0) and the end of the EMDR intervention lasting three months (T1)
  Structural (T1 weigthed 3D and functional MRI (resting state and task activation fMRI)
Expanded Disability Status Scale - EDSS Scale | Change between the baseline (before EMDR treatment-T0), the end of the EMDR intervention lasting three months (T1) and the follow up at three months after the end of the intervention (T2)
  A method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability.

IPD SHARING:
Plan to Share IPD: Undecided